CLINICAL TRIAL: NCT07151768
Title: Prospective Validation of the Novel PVD-B65 Risk Score in Patients With Chronic Lung Disease and Pulmonary Hypertension
Status: Recruiting | Type: Observational
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Other Study IDs: 32278
Record Dates: First submitted 2025-08-12; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lung Disease; Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Observational Study — * assignment of PVD-B65 score derived from standard of care testing
  * no therapeutic intervention or other treatment

SUMMARY:
Prospective observational study to determine if the PVD-B65 risk score for one-year mortality in patients with chronic lung disease and pulmonary hypertension (CLD-PH) can accurately risk stratify these patients and successfully predict one-year mortality from time of pulmonary hypertension diagnosis. PVD-B65 risk score was developed in a retrospective cohort of patients with CLD-PH, utilizing the presence of pulmonary fibrosis without emphysema, pulmonary vascular resistance (PVR) > 5 woods units (WU), 6-minute walk distance (6MWD) < 150 meters, B-natriuretic type peptide (BNP) > 200 pg/mL or N-terminal pro-natriuretic type peptide (NT-proBNP) > 300 pg/dL, and age > 65 years as the score components.

DETAILED DESCRIPTION:
Objectives:

Primary objective: Prospectively validate the PVD-B65 risk score in patients newly diagnosed with or referred to our center with chronic lung disease and pulmonary hypertension by assigning a PVD-B65 score at time of diagnosis and/or referral and following one-year mortality outcome.

Secondary objectives:

* Assess whether the risk severity assigned from the PVD-B65 score in patients newly diagnosed with or referred to our center with chronic lung disease and pulmonary hypertension can predict clinical worsening.
* Assess whether optimal treatment in line with standard of care of both chronic lung disease and pulmonary hypertension can modify the initial risk severity assigned from the PVD-B65 score and in turn influence survival outcomes.

Primary endpoint: One-year outcome of mortality vs. lung transplantation vs. alive without lung transplantation

Secondary endpoints

1. Composite endpoint of clinical worsening defined as hospitalization for respiratory failure, worsening oxygen requirement, intensification of pulmonary vasodilator therapy from initial treatment
2. Change in PH markers (mPAP, PVR, cardiac output, cardiac index via RHC; PASP via TTE, pulmonary artery diameter and pulmonary artery to aorta ratio on CT chest)
3. Change in lung function (FEV1, FVC), 6MWD, and DLCO
4. Change in PVD-B65 score and associated risk severity through duration of study

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria

  1. Adult patients ≥ 18 years of age with chronic lung disease diagnosed via CT chest and/or PFT data and pre-capillary pulmonary hypertension diagnosed via right-heart catheterization (RHC, mPAP > 20 mmHg, PVR > 2 WU, and PCWP ≤ 15 mmHg)

     1. Chronic lung disease diagnoses will include: COPD, IPF, other pulmonary fibrosis, non-fibrotic ILD, combined pulmonary fibrosis and emphysema, and advanced pulmonary sarcoidosis with parenchymal involvement
     2. PFT criteria will include an FEV1/FVC < 0.70 for the diagnosis of COPD
  2. Willingness to make return visits and be available by telephone for the duration of the study.
  3. Ability to participate in necessary testing, including ambulatory testing

Exclusion Criteria:

* Exclusion criteria

  1. Patients with pulmonary hypertension but without associated chronic lung disease (i.e. idiopathic or group 1 PAH, PH with post-capillary component defined as PCWP > 15 mmHg or group 2 PAH, CTEPH or group 4 PH, group 5 PH aside from sarcoidosis with parenchymal involvement)
  2. Patients with uncontrolled severe systemic disease that could influence life expectancy (i.e. uncontrolled cardiovascular disease, active malignancy, etc.)
  3. Prior lung and/or heart transplantation

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic lung disease and pulmonary hypertension
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Prediction of one year mortality | One year
  death (yes or no)

SECONDARY OUTCOMES:
Clinical worsening | one year
  Composite endpoint defined as having had hospitalization for respiratory failure, worsening oxygen requirement in L/min, or intensification of pulmonary vasodilator therapy from initial treatment
Change in PH severity via RHC | Assessed every 6 months for one year
  PVR in Woods units via RHC
Change in PH severity via TTE | Assessed every 3 months for one year
  Estimated PASP in mmHg
Change in functional status | Assessed every 3 months for one year
  6 minute walk distance in meters
Change in PVD-B65 score and associated risk severity through duration of study | Every 3 months for one year
  PVD-B65 risk score (absolute numeric value) calculated throughout study as described above

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States